CLINICAL TRIAL: NCT03811327
Title: Zero-time Exercise for Depression: A Pilot Randomised Controlled Trial
Brief Title: Zero-time Exercise for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY005
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Depression
Keywords: Zero-time Exercise; Depression; Lifestyle; Behavioural Activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Zero-time Exercise group
  Interventions: Behavioral: Zero-time Exercise
- Waitlist group (No Intervention)

INTERVENTIONS:
Behavioral: Zero-time Exercise — A 2-hour group ZTEx training once per week for 2 consecutive weeks (totally 4 hours)
  Arms: Treatment group

SUMMARY:
This study will examine the feasibility and effectiveness of a new lifestyle-integrated exercise, viz. Zero-time Exercise (ZTEx), for the management of depressive symptoms in Chinese adults in Hong Kong. ZTEx refers to the integration of simple strength- and stamina-enhancing physical activity into daily life, which can be done anytime, anywhere and by anyone. Depression is often accompanied by a tendency to sedentary behaviours and sleep disturbances, and sedentary lifestyles is associated with depression. The conventional psychological treatment approach for depression, viz. Cognitive Behavioural Therapy (CBT), emphasises the relationship between activity and mood. One of the treatment components in CBT for depression, viz. Behavioural Activation (BA), aims to promote activity engagement that are reinforcing and consistent with the long-term goals in reducing sedentary behaviour and increasing physical activity. The simple and brief ZTEx uses a foot-in-the-door approach to initiate simple behaviour change as an entry-level step for facilitating BA for participants with depression. A pilot randomized controlled trial (RCT) has shown some evidence on the effectiveness of ZTEx on improving insomnia. However, investigators have found no RCT on the effectiveness of ZTEx for the management of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18-65 years
* Cantonese language fluency
* Patient Health Questionnaire (PHQ-9) score ≥ 10 and ≤ 14; and
* Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

* Pregnancy;
* Have high levels of suicidal ideation (referral information to professional services will be provided);
* Unstable psychotropic drugs within 2 weeks before study entry and throughout the treatment phase;
* Current involvement in psychotherapy for depression;
* Having unsafe conditions and are not recommended for exercising by physicians; and
* Major psychiatric, medical or neurocognitive disorders that would make participation infeasible or interfere with the adherence to physical exercising.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 1-week post-treatment and 4-week post treatment
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline, 1-week post-treatment and 4-week post treatment
  A 14-item self-rating scale that measures anxiety and depression in both hospital and community settings. It is divided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items. It is for screening purpose and not meant to be a diagnostic tool. HADS scores of 8-10, 11-14, and 15-21 represent mild, moderate, and severe anxiety and depression separately
Change in Insomnia Severity Index (ISI) | Baseline, 1-week post-treatment and 4-week post treatment
  A 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem. Total score categories: 0-7 is no clinically significant insomnia, 8-14 is subthreshold insomnia,15-21 is clinical insomnia (moderate severity), and 22-28 is clinical insomnia (severe)
Change in Multidimensional Fatigue Inventory (MFI) | Baseline, 1-week post-treatment and 4-week post treatment
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Scores on each subscale range from 4 to 20, with higher scores indicating greater fatigue
Change in International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, 1-week post-treatment and 4-week post treatment
  IPAQ-C is a short form questionnaire assessing walking, moderate-intensity activities and vigorous-intensity activities undertaken across 4 domains - leisure time physical activity, domestic and gardening (yard) activities, work-related physical activity and transport-related physical activity. Both continuous and categorical scores can be represented. For continuous scoring, the items provide separate scores on the three specific types of activities. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of the three specific type of activities. Median minutes/week or median MET-minutes/week is derived for each type of activity - Walking = 3.3 METs, Moderate PA = 4.0 METs and Vigorous PA = 8.0 METs. For categorical scoring, category 1 represents the lowest level of physical activity, category 2 represents moderate level of physical activity, and category 3 represents the highest level of physical activity.
Change in Short Form (Six-Dimension) Health Survey - The Chinese (Hong Kong) Version (SF-6D) | Baseline, 1-week post-treatment and 4-week post treatment
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state)
Change in Sheehan Disability Scale (SDS) | Baseline, 1-week post-treatment and 4-week post treatment
  A 5-item self-report tool for assessing functional impairment in work/school, social life, and family life. Representation of scores in terms of functional impairment: 0: not at all, 1-3: mildly, 4-6: moderately, 7-9: markedly, 10: extremely
Change in Ecological momentary assessment (EMA) | Baseline, 1-week post-treatment and 4-week post treatment
  A smartphone application will be developed and installed in the participant's smartphones for recording the participants' momentary mood, daytime insomnia symptoms as well as activities.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong